CLINICAL TRIAL: NCT07251465
Title: Effectiveness of Pneumococcal Vaccination (20vPnC) to Prevent All-cause Pneumonia and Lower Respiratory Tract Infections Among Adults ≥18 Years Old With an Increased Risk of Pneumococcal Disease at Kaiser Permanente Southern California.
Brief Title: A Study to Learn How Effective is PCV20 to Help Stop Adults Who Have a Higher Chance of Getting Pneumonia
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: B7471041
Record Dates: First submitted 2025-08-20; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia
Keywords: respiratory tract infections; vaccines
MeSH Terms: conditions — Pneumonia; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — No biospecimens collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults ≥18-64 years old with medical conditions and behavioral risk factors
  Interventions: Biological: Receipt of PCV20
- Adults ≥65 years old
  Interventions: Biological: Receipt of PCV20

INTERVENTIONS:
Biological: Receipt of PCV20 — The main exposure of interest will be receipt of PCV20.

SUMMARY:
The purpose of this study is to learn how effective is PCV20 to help stop adults from getting pneumonia. Pneumonia is an infection of the lungs that can be caused by germs like bacteria, virus, or fungi. This study uses existing healthcare information. No participants will be actively enrolled. The information of participants will be taken from Kaiser Permanente Southern California's (KPSC) electronic health records (EHR).

We will look at the EHR information for adults who meet the following points:

* 18 years of age or older and a KPSC member as of 01 July 2022.
* have been a KPSC member for at least one year before 01 July 2022.
* have not received PCV15.
* have had pneumonia or lower respiratory tract infection within 30 days of 01 July 2022.

The study will begin from 01 July 2022 and will be followed through 30 June 2025. At the end of the follow-up period, the study will compare the number of pneumonia cases among people who receive PCV20 who do not receive it.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years at cohort entry;
2. Continuous enrollment, allowing for 45-day administrative gap, for at least one year prior to cohort entry;
3. At least one outpatient visit in the prior to cohort entry.

Exclusion Criteria:

1. PCV15 received any time before or after the cohort entry date;
2. a diagnosis code in the electronic health record (EHR) for pneumonia or lower respiratory tract infection (LRTI) was made within 30 days prior to cohort entry;
3. Kaiser Permanente Southern California (KPSC) members with zero outpatient visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort consisting of adults ≥18 years who meet eligibility criteria as of 01 July 2022 or who become eligible for the cohort thereafter until the end of the cohort follow-up (30 June 2025) will be classified according to PCV20 exposure and followed until the outcomes of interest, loss to follow-up (i.e., health plan disenrollment or death), or the end of the study period, whichever occurs first. Cohort members will contribute time-segments of unvaccinated or vaccinated follow-up time beginning at the first health care visit after cohort entry for unvaccinated time-segments and at 30-days after PCV20 receipt for vaccinated time segments. During the follow-up period, adults who age into the cohort or who are newly diagnosed with a medical condition recommended for pneumococcal vaccination will be eligible for cohort entry so long as the other eligibility criteria are met.
Sampling Method: Non-Probability Sample
Enrollment: 846279 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
PCV20 vaccine effectiveness (VE) against all-cause pneumonia (ACP) calculated as (1- adjusted hazard ratio [aHR]) × 100% among adults aged ≥18-64 years with medical conditions and behavioral risk factors and among adults ≥65 years old, combined | 3 years
  Estimate overall PCV20 effectiveness against ACP among both adults ≥18-64 years old with medical conditions and behavioral risk factors and among adults ≥65 years old combined

SECONDARY OUTCOMES:
Incidence calculated the number of all-cause pneumonia episodes per 100,000 population among both adults ≥18-64 years old with medical conditions and behavioral risk factors and among adults ≥65 years old combined, and each group separately | 3 years
  Estimate the incidence of all-cause pneumonia by PCV20 vaccination status among both adults ≥18-64 years old with medical conditions and behavioral risk factors and among adults ≥65 years old combined, and each group separately.
Vaccine preventable disease incidence (VPDI) calculated as the difference in incidence rates of all-cause pneumonia for the PCV20 unvaccinated and PCV20 vaccinated groups | 3 years
  Estimate the absolute difference in the incidence of all-cause pneumonia by PCV20 vaccination status among both adults ≥18-64 years old with medical conditions and behavioral risk factors and among adults ≥65 years old combined, and each group separately.
PCV20 VE against ACP calculated as (1-aHR) × 100% separately among adults aged ≥18-64 years with medical conditions and behavioral risk factors and among adults ≥65 years old | 3 years
  Estimate overall PCV20 effectiveness against ACP separately among adults ≥18-64 years old with medical conditions and behavioral risk factors or among adults ≥65 years old

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471041